CLINICAL TRIAL: NCT02484885
Title: Xenon-129 Magnetic Resonance Imaging of Healthy Subjects: Hardware and Software Development and Reproducibility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Grace Parraga, PhD, Scientist. Robarts Research Institute, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ROB0030
Record Dates: First submitted 2015-06-24; First posted 2015-06-30 (Estimated); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Healthy Volunteers
Keywords: Magnetic Resonance Imaging; Pulmonary Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Volunteers (Other): Healthy volunteers will undergo pulmonary function tests, hyperpolarized Xenon MRI at each visit.
  Interventions: Other: Hyperpolarized Xenon MRI

INTERVENTIONS:
Other: Hyperpolarized Xenon MRI — Hyperpolarized noble gas imaging using Xenon-129 has been used to explore structural and functional relationships in the lung in patients with lung disease and healthy controls. In contrast to proton-based MRI imaging, 129Xe gas is used as a contrast agent to directly visualize the airways, and thus ventilation. Whereas the normal density of gas is too low to produce an easily detectable signal, this is overcome by artificially increasing the amount of polarization per unit volume using optical pumping.

SUMMARY:
Healthy volunteers aged 18-85 will undergo hyperpolarized 129-Xe MRI and pulmonary function testing for the development of tools to assess image signal to noise and reproducibility of spin-density and diffusion-weighted imaging.

DETAILED DESCRIPTION:
Briefly, during a one to two hour visit, subjects will provide written informed consent and then undergo: 1) brief medical history and vital signs, 2) full pulmonary function tests, 3) proton MRI, 4) spin-density, diffusion weighted, and/or dissolved phase 129-Xe MRI.

Full pulmonary function tests including spirometry, plethysmography and diffusing capacity of carbon monoxide (DLCO), Multiple Breath Nitrogen Washout (MBNW) to measure Lung Clearance Index (LCI), and Forced Oscillation Technique (FOT) will be performed according to ATS guidelines. MedGraphics Elite Series, MedGraphics Corporation. St. Paul, MN USA and/or nDD EasyOne Spirometer, nDD Medical Technologies Inc. Andover, MA USA will be used. All measurements will be performed in the Pulmonary Function Laboratory at Robarts Research Institute.

Subjects will be placed in the 3T MR scanner with one of three 129-Xe chest coils fitted over their torso and chest. Hearing protection will be provided to each subject to muffle the noise produced by the gradient RF coils. A pulse oximeter lead will be attached to all of the subjects to monitor their heart rate and oxygen saturation. MRI will be performed for up to a period of 30 minutes. All subjects will have supplemental oxygen available via nasal cannula at a flow-rate of 2 liters per minute as a precaution in the event of oxygen desaturation.

ELIGIBILITY:
Inclusion Criteria:

* able to perform a breath hold for up to 16 sec
* BMI between 18 and 40
* stable health on the basis of medical history
* smoking history < 1 pack/year

Exclusion Criteria:

Patient is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material.

* Subject has a daytime room air oxygen saturation <90% while lying supine.
* Patient is unable to perform spirometry or plethysmography maneuvers
* Patient is pregnant
* In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia.
* Subject has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-08; Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Ventilation Defect Percent (VDP) | 5 years

SECONDARY OUTCOMES:
Apparent Diffusion Coefficients (ADC) | 5 years
Dissolved Phase Spectroscopy Measurements | 5 years
  129-Xe dissolved phase MRI data will be reconstructed using a re-gridding method. The following ratios will be determined by the area-under-the curve obtained from spectroscopy: red-blood-cell to alveolar membrane ratio (RBC:membrane); RBC to gas ratio (RBC:gas); and the membrane to gas ratio (membrane:gas). Spectroscopic signals will be used to reconstruct perfusion and alveolar membrane maps.

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario
Locations (1):
- Robarts Research Institute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada